CLINICAL TRIAL: NCT03076918
Title: A Phase II Study Evaluating the Non-inferiority of the Device FLEXITHERALIGHT Compared to the Conventional Photodynamic Therapy (PDT)
Brief Title: Evaluating the Device FLEXITHERALIGHT Compared to the Conventional Photodynamic Therapy
Acronym: Flexithera
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: decision of the investigator in the face of new scientific knowledge
Sponsor: University Hospital, Lille (Other)
Collaborators: National Research Agency, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2013_23; 2013-A01096-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Keratosis, Actinic
Keywords: PDT, Methyl Aminolevulinate, Light Emitting Textile
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: Split face intraindividual comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional PDT (Active Comparator): Aktilite® Galderma
  Interventions: Device: Aktilite® Galderma
- FLEXITHERALIGHT PDT (Experimental): Light Emitting Textile Device
  Interventions: Device: FLEXITHERALIGHT PDT

INTERVENTIONS:
Device: FLEXITHERALIGHT PDT — Preparation of lesions, MAL application+occlusive dressing during 30 minutes+illumination 2.5 hours
  Arms: FLEXITHERALIGHT PDT
Device: Aktilite® Galderma — Preparation of lesions, MAL application+occlusive dressing during 3 hours+illumination 7 to 10 minutes
  Other Names: Conventional PDT
  Arms: Conventional PDT

SUMMARY:
This study compares the efficacy and tolerance of a new device (FLEXITHERALIGHT) for photodynamic therapy in the treatment of keratosis actinic in comparison of classical PDT with Aktilite®.

DETAILED DESCRIPTION:
The study is an intraindividual comparison of two methods. The number of subjects to be enrolled is 47 patients. All participants will receive both two treatments in a single visit : a first period of 2.5 hours of illumination with FLEXITHERALIGHT device followed by a continuous red light Spectrum (between 7 and 10 minutes) with Aktilite® after an appropriate incubation of methyl aminolevulinate).

Patients will complete a pain assessment scale after receiving both treatments, then, 3 follow up visits will be scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of minimum 10 previously untreated not pigmented, non-hyperkeratotic AK lesions of Grade I and II of the forehead and/or scalp (according to Olsen et Al. JAAD 1991, cf. REF 31) where other therapies are unacceptable or considered medically less appropriate with a symmetrical repartition on both side of the forehead and/or scalp. The diagnosis of AK will be determined upon clinical evaluation (i.e. visual inspection and palpation) by the investigator.
* Symmetrical areas in terms of number and severity of lesions. The axis of symmetry between the two areas will be defined by the investigator according to the distribution of lesions.
* The two areas to be treated should not be coalescing. A minimum distance of 10mm is required between the lesions located on the 2 symmetrical areas. A minimum distance of 2 mm is required between the lesions on the same side.
* Minimum 5 lesions with similar dimensions at both symmetrical areas will be treated. If the number of lesions is >7, only 7 lesions on each side will be considered.

Exclusion Criteria:

* Patients with porphyria.
* Patients immunosuppressed for idiopathic, disease specific or therapeutic reasons.
* Use of topical corticosteroids to lesional areas within 2 weeks before PDT.
* Patients receiving local treatment (including cryotherapy and curettage, any - Patients receiving topical treatment (including imiquimod, 5-FU and diclofenac, Picato) in face / scalp area within the last 3 months.
* Use of topical retinoids or alpha-hydroxy acids, urea or systemic retinoids, chemotherapy or immunotherapy within 4 weeks of PDT.
* Pigmented AK lesion(s).
* Known allergy to Metvixia, a similar PDT compound or excipients of the cream including arachis oil, or to peanut or soya.
* Participation in other clinical studies either currently or within the last 30 days.
* Female subjects must be of either:

Non-childbearing potential, i.e. post-menopausal or have a confirmed clinical history of sterility (e.g. the subject is without a uterus) or, Childbearing potential, provided there is a confirmed negative urine pregnancy test prior to study treatment, to rule out pregnancy.

* Any condition which may be associated with a risk of poor protocol compliance.
* Patients currently receiving regular ultraviolet radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Treated lesion response rate | up to month 6
  Each treatment area will be counted, graded with Clinical grade of AK, mapped and photographed

SECONDARY OUTCOMES:
Visual Analog scale of pain | Day 1 and D ay 7.
  Measure the pain and local tolerance graduation range 0 to 10
Scale for clinical assessment of the subject's skin aspect | Months 3 and Months 6
  4-point scale that ranged of Excellent; No scarring, atrophy or induration, and no or slight occurrence of redness or change in pigmentation compared to adjacent skin. Good: No scarring, atrophy or induration but moderate redness or change in pigmentation compared to adjacent skin, Fair: Slight to moderate occurrence of scarring, atrophy or induration, Poor: Extensive occurrence of scarring, atrophy or induration
Fluorescence measure of the PpIX | Baseline, after 3 hours of incubation, in case of treatment interruption, immediately after the treatment, and at 15 and 30 minutes after the end of the treatment.
  Measures with Fluoderm photometer
Irradiance measure in mW/cm2 for each AK | during Aktilite® treatment at Day 1
  Measures realised with a wattmeter OPHIR LaserSTAR to know the power of light delivered
Rate of patients with at least 75% of reduction of the lesions | Months 3 and Months 6
  The reduction in the number of lesions will be calculated as a function of the initial number:≥4 destroyed if 5 lésions; ≥ 5 destroyed if 6 lésions and ≥6 destroyed if 7 lesions
  ≥4 destroyed if 5 lesions
Dermatology Life Quality Index (DLQI) | At Day 7, Months 3 and Months 6
  The questionnaire of 10 questions is completed by the patient to evaluate his quality of life
Satisfaction Questionnaire | At Day 7, Months 3 and Months 6
  The questionnaire es created by the investigator to evaluate the comfort of the device. Patient will give his overall satisfaction and the will answer 7 questions on a 5-point scale that ranged from Not embarrassing, few embarrassing, embarrassing, Very embarrassing, I Don't know

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mortier, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lecomte F, Vignion-Dewalle AS, Vicentini C, Thecua E, Deleporte P, Duhamel A, Mordon S, Mortier L. Evaluating the Noninferiority of a New Photodynamic Therapy (Flexitheralight) Compared With Conventional Treatment for Actinic Keratosis: Protocol for a Phase 2 Study. JMIR Res Protoc. 2019 Apr 26;8(4):e11530. doi: 10.2196/11530. PMID 31025952